CLINICAL TRIAL: NCT03948503
Title: Mulligan Concept in the Treatment of Subacute Ankle Sprains: a Randomized Placebo Trial.
Brief Title: Mulligan Concept in the Treatment of Ankle Sprains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/21NOV/439
Record Dates: First submitted 2019-03-19; First posted 2019-05-14 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Ankle Sprain 1St Degree; Ankle Sprain 2Nd Degree
Keywords: ankle sprain; Mulligan; manual therapy
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with movement (MWM) group (Experimental): Application of the Mulligan concept
  Interventions: Procedure: Mulligan concept
- Sham group (Placebo Comparator): Sham treatment
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Mulligan concept — Mobilization with movement during an active dorsi-flexion of the ankle
  Arms: Mobilization with movement (MWM) group
Procedure: Placebo — Sham mobilization with movement during an active dorsi-flexion of the ankle
  Arms: Sham group

SUMMARY:
Aim of the study is to establish the efficiency of the mulligan concept vs a sham group (who will also serve as control). Patient with an subacute ankle sprains will be assess following the mulligan concept and then randomized in two groups: Mobilization with movement (MWM) group and Sham group. MWM group will receive 3 sets of 10 repetitions of treatment (i.e. passive accessory glide during an active dorsiflexion) while the sham treatment will do 3 sets of 10 active dorsiflexion with the hand of the Physiotherapist only apply on the skin. 3 sessions with 4 days apart will take place. outcomes will be measure before and after every sessions.

DETAILED DESCRIPTION:
All included subject will received the Mulligan concept assessment. First investigator will applied non-weight bearing inferior tibiofibular mobilization with movement (MWM), i.e. passive accessory glide in a posterior and superior direction on the inferior tibiofibular joint. If not painful, Weightbearing inferior tibiofibular MWM will be applied 6 times. it consist on applying a passive accessory glide on the subject while he/she is doing an active dorsiflexion of the injured ankle. Dorsiflexion range of motion, pain and function will be reassess. If either one of previously cited outcomes is improve, subject is considered respondents. If he/she feels any pain or no improvements at all, he/she will be considered non-respondents. If non-weight-bearing inferior tibiofibular MWM is painful, talocrural MWM will be apply, first in non-weightbearing and if painfree, in weight bearing position. Talocrural MWM consist on a posterior glide of the talus while the subject realized an active dorsiflexion of the injured ankle. Same outcomes as previsouly cited will be assess and will determine if the patient is respondent or non-respondent. If the subject is non-respondent of the talocrural MWM or if he/she felt any pain during the talocrural MWM, a non weightbearing cubometatarsal MWM, i.e. cranio-caudal glide of the lateral cubometatarsal joint during an active dorsiflexion of the injured ankle, will be applied. If painfree, a tape will be placed as to replicate the cubometatarsal MWM, and the patient will reassess ROM, pain and function with the tape to see whether he/she is a respondent or non respondent subject. If the subject is non-respondent to neither of the three MWM, he/she is considered a drop-out. Respondent patient will then be randomized into two groups: MWM group and Sham group. MWM group will receive 3 sessions with 4 days apart of 3 sets of 10 repetitions of preferential MWM (inferior tibiofibular, talocrural, cubometatarsal) while the sham group will receive 3 sessions with 4 days apart of 3 sets of 10 repetitions with the first investigator doing a light touch during an active dorsiflexion, mimicking the real MWM techniques. Outcomes will be measures at T0 (beginning of the treatment-beginning of the first session), T1 (end of the first session), T2 (beginning of the second session), T3 (end of the second session), T4 (beginning of the third session) and T5 (end of the treatment-end of the third session).

ELIGIBILITY:
Inclusion Criteria:

* ankle sprain since 2 weeks to 12 weeks
* Grade 1 or 2 ankle sprain
* Asymetrical dorsi-flexion limitation

Exclusion Criteria:

* Acute or Grade 3 ankle sprain
* More than 12 weeks ankle sprain
* Any other trauma of the lower limb

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Ankle dorsiflexion Range of motion | At the beginning (Time1) and end (Time2) of each session (one session is 30 minutes). Every session is separated by 4 days. Outcomes is taken at Day 1(session1) at Time1 & Time2 ,Day 5(session2) at Time1 & Time2 and Day 9(session3) at Time1 & Time2 .
  Wall toe test (distance in cm and degree in °)

SECONDARY OUTCOMES:
Change in Pain | At the beginning (Time1) and end (Time2) of each session (one session is 30 minutes). Every session is separated by 4 days. Outcomes is taken at Day 1(session1) at Time1 & Time2 ,Day 5(session2) at Time1 & Time2 and Day 9(session3) at Time1 & Time2 .
  a 10cm Visual Analog Scale
Change in Stiffness sensation | At the beginning (Time1) and end (Time2) of each session (one session is 30 minutes). Every session is separated by 4 days. Outcomes is taken at Day 1(session1) at Time1 & Time2 ,Day 5(session2) at Time1 & Time2 and Day 9(session3) at Time1 & Time2 .
  Visual Analog Scale (VAS)
Change in Dynamic function | At the beginning (Time1) and end (Time2) of each session (one session is 30 minutes). Every session is separated by 4 days. Outcomes is taken at Day 1(session1) at Time1 & Time2 ,Day 5(session2) at Time1 & Time2 and Day 9(session3) at Time1 & Time2 .
  Y-test
Change in fonctionnel movement | At the beginning (Time1) of Day1 (Session1) and end of Day9 (Session3). One session is 30 minutes long. Each session is separated by 4 days.
  Forward step down test
Change inDaily-life function | At the beginning (Time1) of Day1 (Session1) and end (Time2) of Day9 (Session3). One session is 30 minutes long. Each session is separated by 4 days.
  Foot and Ankle Ability Measure (FAAM) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Mahaudens, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No